CLINICAL TRIAL: NCT06836284
Title: Evaluation of a Digital Treatment Tool in Combination With Anti-Obesity Medications
Brief Title: The Evira Study: Additional Support During Anti-Obesity Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Evira AB (Industry)
Responsible Party: Principal Investigator, Pernilla Danielsson, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-07214-01
Record Dates: First submitted 2025-01-29; First posted 2025-02-20 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Childhood Obesity; Treatment Adherence
Keywords: Mobile Health; Self-Monitoring; Digital Treatment; Anti-Obesity Medication
MeSH Terms: conditions — Pediatric Obesity; Treatment Adherence and Compliance | interventions — Liraglutide; semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anti-obesity medication liraglutide or semaglutide combined with digi-physical treatment Evira (Active Comparator): Patients randomized to this group will receive liraglutide or semaglutide in combination with a digi-physical treatment tool, named Evira. Patients will be provided with a digitless measuring scale intended for daily use at home. They will be able to communicate with clinical staff at pivotal moments.
  Interventions: Device: Digi-physical treatment tool, Evira; Drug: Anti-obesity medication with liraglutide or semaglutide
- Control group (Other): Patients randomized to this group will receive liraglutide or semaglutide treatment according to the clinic's standard procedures.
  Interventions: Drug: Anti-obesity medication with liraglutide or semaglutide

INTERVENTIONS:
Device: Digi-physical treatment tool, Evira — A digi-physical treatment tool named Evira will be used to provide behavioral treatment.
  Arms: Anti-obesity medication liraglutide or semaglutide combined with digi-physical treatment Evira
Drug: Anti-obesity medication with liraglutide or semaglutide — Anti-obesity medication with liraglutide or semaglutide according to the clinic's standard procedure

SUMMARY:
The goal of this clinical trial is to evaluate the effect of adding a digi-physical treatment tool as a complement to the local treatment with anti-obesity medication in adolescents with obesity. The main question it aims to answer is:

- Can a combination of a digi-physical treatment tool and anti-obesity medication improve treatment outcomes for patients with obesity compared to patients treated with anti-obesity medications alone?

This is a randomized controlled two-arm multicenter study where participants will be randomized to the intervention group (digi-physical treatment+medication) or control group (medication only). Participants will be followed for six months.

DETAILED DESCRIPTION:
Obesity is a complex and multifactorial disease, highlighting the need to develop treatment strategies that achieve more sustainable and effective outcomes. Treatments with the medications liraglutide and semaglutide have been tested, showing effects of -0.23 and -1.10 BMI SDS units, respectively, after approximately one year in individuals aged 12-17 years. These results are significantly better than those achieved with conventional treatment, where the effect for adolescents over 12 years is close to zero. However, long-term results indicate that many patients, after discontinuing medication, quickly return to the same degree of obesity they had at the start of the study.

Anti-obesity medications can be effective for many patients, but challenges remain in achieving better treatment outcomes for more individuals. This underscores the need to evaluate whether the effect can be optimized by combining medication with digital treatment tools.

Evira is a digital treatment tool that enables close monitoring of objective treatment outcomes and continuous communication between healthcare professionals and families. The tool includes daily measurements conducted in the home of the patient on a measuring device that do not display any numbers. The device is linked to a mobile app where weight trends are displayed as a moving average in the form of BMI standard deviation score (BMI SDS). The app also provides an individualized target curve, visualizing the expected weight trajectory. Since weight changes in growing children are complex to interpret, BMI SDS is used as a standard metric. Objective data from the measuring device are also automatically transmitted to a clinic interface, enabling direct communication between the clinic and the family via the app.

This study is a randomized controlled two-arm multicenter trial conducted across multiple centers in Sweden that use liraglutide and semaglutide. Patients will be randomized in a 2:1 ratio, with two-thirds allocated to the intervention group and receiving medications combined with the Evira digital treatment tool, and one-third allocated to the control group, receiving medications with standard clinic support. Patients will be followed for six months. Data collection will include physical examinations, background information, and electronically distributed questionnaires administered to both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients offered liraglutide or semaglutide in accordance with the clinic's routines.
* Aged 12-17 years at the time of inclusion.
* The family agrees to participate in a clinical study.

Exclusion Criteria:

* Endocrine disorders other than well-controlled hypothyroidism.
* Severe neuropsychiatric disorders that may affect adherence to the study.
* Eating disorder requiring treatment within the last six months before inclusion or observed during screening prior to inclusion.
* Somatic conditions that may complicate the evaluation of treatment outcomes, such as patients on irregular oral corticosteroid treatment.
* Hypothalamic or monogenic obesity, and genetic syndromes such as Down syndrome.
* Patients deemed unsuitable for participation by the responsible physician.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-10-07 (Estimated); Primary Completion 2026-08-29 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in BMI SDS | From start of treatment to six months follow-up
  Weight and height will be combined to report BMI in kg/m^2 for analyzing change in BMI standard deviation score.

SECONDARY OUTCOMES:
Proportion achieving less favorable reduction in BMI SDS | From start of treatment to six months follow-up
  Can the proportion of patients achieving less favorable outcomes than those reported in published studies (liraglutide BMI SDS reduction of -0.23 units, semaglutide BMI SDS reduction of -0.75 units after six months) be reduced by combining medication treatment with a digital treatment tool?
Treatment Adherence | From start of treatment to six months follow-up
  What is the treatment effect in relation to compliance based on the number of home measurements, physical visits, and in-app messages in the intervention group?
Side effects | From start of treatment to six months follow-up
  What is the incidence of potential side effects and treatment discontinuation?
Professionals perception of the digital tool | From start of treatment to six months follow-up
  Questionnaires regarding how healthcare professionals perceive the use of the digital tool in combination with medication treatment including questions such as; does it facilitate your work? Does it take more or less time? (Evira specific questionnaire)
Patients perception of the treatment and digital tool | From start of treatment to six months follow-up
  Questionnaire regarding how patients perceive the treatment and support received during the study, including questions such as; did you get enough and timely support from your healthcare provider? (Evira constructed questionnaire)
Patients Quality of life | From start of treatment to six months follow-up
  How do patients rate their quality of life before, during, and after the study period? Are there differences between the intervention and control groups?
  PROMIS version Pediatric-25 Profile GenPop v3.0 will be used. The instrument contains six domains (see below) along with a single item on Pain Intensity (scoring 0-10, 0=no pain, 10=worst pain).
  T-scores are used to assess the health domains, a T-score of 50 represents the average with a standard deviation of 10.
  For negatively-worded domains (Anxiety, Depressive Symptoms, Fatigue and Pain Interference), higher T-scores indicate worse health status.
  For positively-worded domains (Physical Function-Mobility and Peer Relationships), higher T-scores indicate better health status.

CONTACTS AND LOCATIONS:
Locations (1):
- HKH Crown Princess Victoria's Childrens and youth Hospital Linköping, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Undecided